CLINICAL TRIAL: NCT03686514
Title: The Impact of Imprinting and Repeated Influenza Vaccination on Adaptive Immunity, Transcriptomics, and Metabolomics
Acronym: FLU2
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study closed prior to completing year 3 of the study due to the COVID-19 pandemic.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Nadine Rouphael, Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00106407
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Results first posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-06

CONDITIONS: Influenza
Keywords: Flu vaccine; Influenza vaccine; Immune response; Influenza strain
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- H3N2 birth cohort (Experimental): The H3N2 cohort consists of participants born between 1968-1977.
  Interventions: Biological: FLUARIX QUADRIVALENT
- H1N1 birth cohort (Experimental): The H1N1 cohort consists of participants born between 1948-1957.
  Interventions: Biological: FLUARIX QUADRIVALENT

INTERVENTIONS:
Biological: FLUARIX QUADRIVALENT — The FDA-approved, quadrivalent seasonal influenza vaccine that will be administered contains four distinct strains, two influenza A viruses and two influenza B viruses.

SUMMARY:
The goal of this study is to understand the impact on the human immune system's response to the four strain flu vaccine in individuals who have "imprinted" on specific influenza strains. It will also consider the effects of repeated prior annual influenza vaccination on the immune system.

DETAILED DESCRIPTION:
Seasonal influenza outbreaks continue to cause substantial disease burden, with an estimated 3-5 million cases of severe illness, and 250,000 to 500,000 deaths worldwide each year. In the United States, the Centers for Disease Control and Prevention (CDC) reports that influenza has resulted in 9.2-35.6 million illnesses with 12,000-56,000 deaths annually since 2010. There is an urgent need to better understand the immunologic responses to current licensed vaccines in order to develop a more effective vaccine that does not rely on annual updates, provides broad protection, and is durable; i.e., a universal influenza vaccine.

The immune response to the influenza vaccine is affected by many parameters, including prior imprinting to a specific influenza strain based on birth cohort, as well as prior influenza vaccination. The FDA-approved, quadrivalent seasonal influenza vaccine that will be administered contains four distinct strains, two influenza A viruses (IAVs) and two influenza B viruses (IBVs). The approved seasonal influenza vaccine will be given for each season of influenza: 2018-2019, 2019-2020, and 2020-2021.

This study is a prospective pilot study conducted over the course of three years (with three specific influenza seasons studied). For each year (2018-2019, 2019-2020, and 2020-2021), two cohorts of 10 participants each, who are in good health and meet all eligibility criteria, will be recruited. The influenza A virus subtype H3N2 cohort (N=30 total, 10 per year) will consist of participants born between 1968-1977, and the influenza A virus subtype H1N1 cohort (N=30 total, 10 per year) will consist of participants born between 1948-1957. Each participant will make a total of six visits to the Hope Clinic. Day 1 will include the informed consent process, and screening to ensure the subject meets all inclusion criteria and meets no exclusion criteria. For the consenting and eligible subject, the visit will also include pre-vaccination phlebotomy for baseline immunogenicity laboratory assays. After baseline sample collection, the participants will receive the FDA-approved seasonal influenza vaccine. Subsequent study visits up to 180 days post-vaccination will include collection for immunogenicity assays.

This study is not powered to test a formal null hypothesis. Rather, it is a hypothesis-generating investigation that will hopefully lead to larger trials based on the findings. The study will be conducted over the course of three years to increase the total sample population size and to validate the findings over different influenza seasons.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of informed consent and provision of written informed consent before any study procedures.
2. Capable of attending all study visits according to the study schedule.
3. Males or females born between 1968-1977 or 1948-1957.
4. Are in good health, as determined by medical history and targeted physical exam related to this history.
5. Oral temperature is less than 38 degrees Celsius.
6. Resting pulse rate is between 50 and 100 beats per minute.
7. Female subjects of childbearing age must have a negative urine pregnancy test within 24 hours before study vaccination.
8. Have received the influenza vaccine at least 3 of the past 5 years or have received the influenza vaccine in 2 or less of the past 5 years.

Exclusion Criteria:

1. Have an acute illness within 72 hours before vaccination.
2. Have any condition that, in the opinion of the principal investigator, would place the subject at an unacceptable risk of harm or confound the interpretation of the study results.
3. Have any acute or chronic medical condition that, in the opinion of the principal investigator, would make vaccination unsafe or interfere with the evaluation of immune response to study vaccination.
4. Have a suppressed immune system as a result of illness, immunosuppressive medication, chemotherapy, or radiation therapy within 3 years prior to study vaccination.
5. Have known HIV, hepatitis B, or hepatitis C infection.
6. Have a known history of autoimmune disease.
7. Have taken oral or parenteral corticosteroids of any dose within 30 days before study vaccination.
8. Have taken high-dose inhaled corticosteroids within 30 days before study vaccination.
9. Have received, or plan to receive, any licensed live vaccine within 30 days, or any licensed inactivated vaccine within 14 days, prior to, or after, study vaccination.
10. Have planned receipt of any unlicensed or investigational medications, biologics, or vaccines for the duration of subject study participation.
11. Have received immunoglobulin or other blood products, with the exception of Rho D immunoglobulin, within 90 days prior to study vaccination.
12. Have donated blood or blood products within 30 days before study vaccination, or within 60 days after study vaccination, or plan to donate blood within 30 days of the last blood draw.
13. Have known hypersensitivity or allergy to eggs, egg protein, chicken protein, or other compounds of the study vaccine.
14. Have a history of severe reactions following vaccination with influenza virus vaccines.

Ages: 42 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Rouphael, MD, Principal Investigator — Emory University
Locations (1):
- The Hope Clinic of the Emory Vaccine Center, Atlanta, Georgia, United States

REFERENCES:
- [Result] Sherman AC, Lai L, Bower M, Natrajan MS, Huerta C, Karmali V, Kleinhenz J, Xu Y, Rouphael N, Mulligan MJ. The Effects of Imprinting and Repeated Seasonal Influenza Vaccination on Adaptive Immunity after Influenza Vaccination. Vaccines (Basel). 2020 Nov 7;8(4):663. doi: 10.3390/vaccines8040663. PMID 33171854

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant enrollment began October 22, 2018 and all follow up was complete by June 20, 2020. Participants were enrolled at the Hope Clinic of the Emory Vaccine Center in Atlanta, Georgia, USA.
Pre-assignment Details: Individuals were permitted to participate in multiple years of the study. One individual belonging to the H1N1 Birth Cohort, born between the years of 1948 and 1957, participated in both the 2018-2019 and 2019-2020 vaccine years. Thus, each vaccine year for this cohort had 10 participants, but there were 19 discrete individuals overall.
Groups:
- H3N2 Birth Cohort, Born Between 1968 and 1977: The H3N2 cohort consists of participants who were born between 1968-1977. Participants received the FLUARIX QUADRIVALENT flu vaccine for the 2018-2019 vaccine year or the 2019-2020 vaccine year. The FDA-approved, quadrivalent seasonal influenza vaccine administered contained four distinct strains, two influenza A viruses and two influenza B viruses.
- H1N1 Birth Cohort, Born Between 1948 and 1957: The H1N1 cohort consists of participants who were born between 1948-1957. Participants received the FLUARIX QUADRIVALENT flu vaccine for the 2018-2019 vaccine year and/or the 2019-2020 vaccine year. The FDA-approved, quadrivalent seasonal influenza vaccine administered contained four distinct strains, two influenza A viruses and two influenza B viruses.
Period: Overall Study
Arm/Group | H3N2 Birth Cohort, Born Between 1968 and 1977 | H1N1 Birth Cohort, Born Between 1948 and 1957
Started | 20 | 19
Started 2018-2019 Vaccine Year | 10 | 10
Completed 2018-2019 Vaccine Follow up | 10 | 10
Started 2019-2020 Vaccine Year | 10 | 10
Completed 2019-2020 Vaccine Follow up | 10 | 10
Completed | 20 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | H3N2 Birth Cohort, Born Between 1968 and 1977 | H1N1 Birth Cohort, Born Between 1948 and 1957 | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 7 | 27
  >=65 years | 0 | 12 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.39 (2.77) | 66.95 (2.29) | 55.89 (11.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 11 | 8 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 19 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 11 | 16 | 27
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Achieving Seroprotection Against Each Strain
Description: Seroprotection against each strain contained in the seasonal quadrivalent influenza vaccine (A/H1N1, A/H3N2, B/Phuket, and B/Colorado) were measured by hemagglutination inhibition (HAI) antibody response. Seroprotection is defined as a titer of ≥ 40.
Time Frame: 28 days after vaccination
Population: The data for the individual in the H1N1 Birth Cohort who participated in both vaccine years is included for each year of participation.
Measure: Count of Participants; unit: Participants
Arm/Group | H3N2 Birth Cohort, Born Between 1968 and 1977 | H1N1 Birth Cohort, Born Between 1948 and 1957
Number analyzed (Participants) | 20 | 20
Participants
  A/H1N1 | 19 | 20
  A/H3N2 | 20 | 17
  B/Phuket | 19 | 17
  B/Colorado | 20 | 20

2. Primary Outcome: The Number of Participants Achieving Seroconversion Against Each Strain
Description: Seroconversion against each strain contained in the seasonal quadrivalent influenza vaccine was measured by HAI antibody response. Seroconversion is defined as a four-fold rise in HAI post- compared to pre-vaccination, or a titer of ≥40 if the pre-vaccination titer was <10.
Time Frame: 28 days after vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | H3N2 Birth Cohort, Born Between 1968 and 1977 | H1N1 Birth Cohort, Born Between 1948 and 1957
Number analyzed (Participants) | 20 | 20
Participants
  A/H1N1 | 11 | 10
  A/H3N2 | 12 | 10
  B/Phuket | 9 | 11
  B/Colorado | 8 | 8

3. Primary Outcome: Geometric Mean Titers (GMTs) of Serum HAI Against Each Strain
Description: The geometric scale is logarithmic. A geometric mean is calculated by averaging the logarithms of the test values and then converting the mean to a real number.
Time Frame: 28 days after vaccination
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: GMTs
Arm/Group | H3N2 Birth Cohort, Born Between 1968 and 1977 | H1N1 Birth Cohort, Born Between 1948 and 1957
Number analyzed (Participants) | 20 | 20
GMTs
  A/H1N1 | 282.5 (301) | 389 (575)
  A/H3N2 | 458 (564) | 539 (1097)
  B/Phuket | 463 (579) | 200 (183)
  B/Colorado | 258 (273) | 180 (260)

4. Secondary Outcome: The Proportion of Participants Achieving Seroprotection or Seroconversion Against Each Strain Measured by Neutralizing Antibody (NAb) Response
Description: Seroprotection/seroconversion against each strain contained in the seasonal quadrivalent influenza vaccine will be measured by neutralizing antibody (NAb) response. The proportion of subjects achieving seroprotection (titer of ≥ 40) or seroconversion (four-fold rise in NAb post- compared to pre-vaccination, or a titer of ≥40 if the pre-vaccination titer was <10) against each strain will be assessed.
Time Frame: 28 days after vaccination
Population: NAb testing was not performed as all research efforts moved to coronavirus disease 2019 (COVID-19) research.
Arm/Group | H3N2 Birth Cohort, Born Between 1968 and 1977 | H1N1 Birth Cohort, Born Between 1948 and 1957
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum NAb Against Each Strain
Description: as for outcome 3
Time Frame: 28 days after vaccination
Population: NAb testing was not performed as all research efforts moved to COVID-19 research.
Arm/Group | H3N2 Birth Cohort, Born Between 1968 and 1977 | H1N1 Birth Cohort, Born Between 1948 and 1957
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: The Number of Participants Achieving Seroprotection Against Each Strain
Description: as for outcome 1
Time Frame: 180 days after vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | H3N2 Birth Cohort, Born Between 1968 and 1977 | H1N1 Birth Cohort, Born Between 1948 and 1957
Number analyzed (Participants) | 20 | 20
Participants
  A/H1N1 | 18 | 17
  A/H3N2 | 17 | 12
  B/Phuket | 17 | 14
  B/Colorado | 18 | 20

7. Secondary Outcome: The Number of Participants Achieving Seroconversion Against Each Strain
Description: as for outcome 2
Time Frame: 180 days after vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | H3N2 Birth Cohort, Born Between 1968 and 1977 | H1N1 Birth Cohort, Born Between 1948 and 1957
Number analyzed (Participants) | 20 | 20
Participants
  A/H1N1 | 7 | 7
  A/H3N2 | 5 | 6
  B/Phuket | 4 | 5
  B/Colorado | 3 | 7

8. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum HAI Against Each Strain
Description: as for outcome 3
Time Frame: 180 days after vaccination
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: GMTs
Arm/Group | H3N2 Birth Cohort, Born Between 1968 and 1977 | H1N1 Birth Cohort, Born Between 1948 and 1957
Number analyzed (Participants) | 20 | 20
GMTs
  A/H1N1 | 151.2 (153) | 197 (191)
  A/H3N2 | 124 (147) | 185 (297)
  B/Phuket | 135 (112) | 114 (92)
  B/Colorado | 130 (157) | 98 (67)

9. Secondary Outcome: The Proportion of Participants Achieving Seroprotection or Seroconversion Against Each Strain Measured by NAb Response
Description: Seroprotection/seroconversion against each strain contained in the seasonal quadrivalent influenza vaccine will be measured by NAb antibody response.
Time Frame: 180 days after vaccination
Population: NAb testing was not performed as all research efforts moved to COVID-19 research.
Arm/Group | H3N2 Birth Cohort, Born Between 1968 and 1977 | H1N1 Birth Cohort, Born Between 1948 and 1957
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum NAb Against Each Strain
Description: as for outcome 3
Time Frame: 180 days after vaccination
Population: NAb testing was not performed as all research efforts moved to COVID-19 research.
Arm/Group | H3N2 Birth Cohort, Born Between 1968 and 1977 | H1N1 Birth Cohort, Born Between 1948 and 1957
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning during the first study visit when the influenza vaccine was administered through the final study assessment at 180 days post-vaccination.
Groups:
- H1N1 Birth Cohort, Born Between 1948 and 1957: The H1N1 cohort consists of participants who were born between 1948-1957. Participants received the FLUARIX QUADRIVALENT flu vaccine for the 2018-2019 vaccine year and/or the 2019-2020 vaccine year. The FDA-approved, quadrivalent seasonal influenza vaccine administered contained four distinct strains, two influenza A viruses and two influenza B viruses. One individual participated in both vaccine years and is counted only once for adverse event reporting.
Arm/Group | H3N2 Birth Cohort, Born Between 1968 and 1977 | H1N1 Birth Cohort, Born Between 1948 and 1957
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19

LIMITATIONS AND CAVEATS:
Due to the COVID-19 pandemic, this study was terminated prior to beginning year 3 of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-13): https://cdn.clinicaltrials.gov/large-docs/14/NCT03686514/Prot_SAP_000.pdf